CLINICAL TRIAL: NCT02558127
Title: Asthma With Hypersecretion-associated Gene for Cystic Fibrosis Clinical, Inflammatory and Genetics Characterization
Brief Title: Asthma With Hypersecretion-associated Gene for Cystic Fibrosis
Acronym: CF-asthma
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-CFT-2014-68; ESR-15-10784 (Registry Identifier: AstraZeneca)
Record Dates: First submitted 2015-06-15; First posted 2015-09-23 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-02

CONDITIONS: Asthma
Keywords: asthma; cystic fibrosis
MeSH Terms: conditions — Asthma; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — From peripheral blood samples, the DNA extraction following the protocol saline method. From the DNA samples obtained CFTR gene analysis to detect genetic variants by sequencing or mass Next Generation Sequencing (NGS) in Miseq team Illumina platform (available in the Hospital de la Santa Creu i Sant be held Pau).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 50 asthma patients: 50 asthma patients with bronchial mucus hypersecretion
  Interventions: Genetic: Asthma patients
- asthma patients: 50 asthma patients without bronchial mucus hypersecretion
  Interventions: Genetic: Asthma patients

INTERVENTIONS:
Genetic: Asthma patients — Patients with inclusion criteria, following examinations: a study of lung function measurement of the fraction of nitric oxide in exhaled air, induced sputum, sputum, and extraction of peripheral venous blood for Study of genetic variants in the CFTR gene,skin prick test . The number of eosinophils in peripheral blood by automated cell counting and Total IgE by ELISA were measured. Furthermore, the level of asthma control be assessed by validated symptom questionnaire Asthma Control Test, quality of life is determined by the MiniAQLQ questionnaire.

SUMMARY:
The combination of asthma and being a carrier of genetic variants (mutations and / or polymorphisms) in the CFTR gene variant would cause bronchial asthma with mucus hypersecretion. This phenotype is characterized by a more severe disease, in terms of control, quality of life, exacerbations and lung function, and a different asthma the bronchial hypersecretion without inflammatory phenotype.

DETAILED DESCRIPTION:
Primary objective:

Determine the presence of genetic variants (mutations and / or polymorphisms) of the CFTR gene in patients with asthma with or without bronchial mucus hypersecretion.

Secondary objectives:

To identify genetic variants (mutations and / or polymorphisms) of the most common CFTR gene in the asthmatic population. -To define the inflammatory phenotype of asthma with bronchial mucus hypersecretion. -To compare the severity, control, quality of life and frequency of exacerbations of asthma patients with or without bronchial mucus hypersecretion

ELIGIBILITY:
Inclusion criteria: Asthmatic patients aged between 18 and 80 years.They have not a respiratory infection in the last month.

Criteria for exclusion: Presence of other lung disease, Sequelae of tuberculosis, Bronchiectasis (large, secondary to a different asthma respiratory disease), Cystic fibrosis, Residual pleural disease, Interstitial diseases, Severe comorbidity, Patients with oral corticosteroids or other immunomodulators by causes other than asthma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 100 asthmatic patients of both sexes, aged between 18 and 80 years will be included in the study. They have not a respiratory infection in the last month. Of the 100 patients, 50 will be hypersecretory asthmatic patients and 50 non- hypersecretory asthmatic patients. Both groups have an even distribution regarding sex, age, level and disease control. Asthma patients were defined according to the criteria of the GEMA 2015 -GINA 2014
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of asthmatic patients CF carriers | 12 months

SECONDARY OUTCOMES:
Noncarriers number of asthmatics | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Crespo, Principal Investigator — Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau - IIB Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau. Carrer Mas Casanovas 90., Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goodwin J, Spitale N, Yaghi A, Dolovich M, Nair P. Cystic fibrosis transmembrane conductance regulator gene abnormalities in patients with asthma and recurrent neutrophilic bronchitis. Can Respir J. 2012 Jan-Feb;19(1):46-8. doi: 10.1155/2012/546702. PMID 22332135
- [Result] Dahl M, Tybjaerg-Hansen A, Lange P, Nordestgaard BG. DeltaF508 heterozygosity in cystic fibrosis and susceptibility to asthma. Lancet. 1998 Jun 27;351(9120):1911-3. doi: 10.1016/s0140-6736(97)11419-2. PMID 9654257
- [Result] Dahl M, Nordestgaard BG, Lange P, Tybjaerg-Hansen A. Fifteen-year follow-up of pulmonary function in individuals heterozygous for the cystic fibrosis phenylalanine-508 deletion. J Allergy Clin Immunol. 2001 May;107(5):818-23. doi: 10.1067/mai.2001.114117. PMID 11344348